CLINICAL TRIAL: NCT05779865
Title: Study of Different Gating Techniques of Positron Emission Tomography Acquisition Focus on Lung or Liver Nodules. Comparaison on Phantoms and a Series of Patients
Brief Title: Study of Different Gating Techniques for PET Image of Lung and Liver Lesions
Acronym: PETGATQUANT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: 23-04
Record Dates: First submitted 2023-02-09; First posted 2023-03-22 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Lung; Nodule; Liver Metastases
Keywords: positron emission tomography; nodule uptake; gating; quantification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lesions blurred by respiratory motion are common in fluorine-18 PET/CT studies. To avoid these artefacts, several standard gating correction technics are available. the investigator aimed to compare the impact of different gating techniques based on phase, amplitude, elastic-motion monitored with and without pressurre sensor device on standardized uptake value (SUVmax and SUVpeak) and uptake volume (UV) measurements on different sizes of pulmonary and liver lesions. The feasability of this study will be done using anthropomorphic coupled with a motion phantom and on a series of patients.

DETAILED DESCRIPTION:
PET-CT images will be acquired on a Biograph Vision600 PET/CT, fitted with 26cm axial field of view and time of flight.

Phantom study will use an anthropomorphic TORSO phantom with a programmable motion phantom, mimicking respiratory motion (QUASAR). Spheres with various internal diameters will be introduce into the lungs (air density) adding an axial mechanical device simulating breathing movement of +/-20mm. Concentration in the spheres will be the same for all diameters. The background and liver activities will be approximatively respectively 38 and 14 MBq. This phantom will be a simulating patient only for lung lesions.

The investigator will compare 6 different PET acquisitions: standard 3min acquisition without movement as our reference of "trues SUVmax and UV", 3min acquisition with simulated breathing movement without any gating and 3min with respectively gating techniques based on phase, amplitude, elastic-motion monitored with and without pressurre sensor device.

Patient study will be on 50 consecutive patients with lung or liver nodules. 18F-FDG injection will be around 2.5 MBq/kg.

The investigator will compare 5 different PET acquisitions: standard acquisition with free respiratory movement as our reference of "trues SUVmax and UV", acquisitions with respectively gating techniques based on phase, amplitude, elastic-motion monitored with and without pressurre sensor device.

ELIGIBILITY:
Inclusion Criteria:

* presence at least of one hepatic or lung nodule

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung or liver nodules
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Comparison of the different gating systems in lung lesions visualization | Inclusion
  Classification, based on a phantom and patients studies, of the different gating system in view of the volume and SUV (max and peak) modification for lung lesions

SECONDARY OUTCOMES:
Comparison of the different gating systems in liver lesions visualization | Inclusion
  Classification, based on a patients studies, of the different gating system in view of the volume and SUV (max and peak) modification for liver lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

REFERENCES:
- [Background] Meier JG, Wu CC, Betancourt Cuellar SL, Truong MT, Erasmus JR, Einstein S, Mawlawi O. Evaluation of a novel elastic respiratory motion correction algorithm on quantification and image quality in abdomino-thoracic PET/CT. J Nucl Med. 2018 Aug 16;60(2):279-284. doi: 10.2967/jnumed.118.213884. Online ahead of print. PMID 30115689
- [Background] Soret M, Bacharach SL, Buvat I. Partial-volume effect in PET tumor imaging. J Nucl Med. 2007 Jun;48(6):932-45. doi: 10.2967/jnumed.106.035774. Epub 2007 May 15. PMID 17504879